CLINICAL TRIAL: NCT04725045
Title: Investigating the Use of Complex Pulse Shapes for DBS in Movement Disorders
Acronym: INSHAPE_DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Myles Mc Laughlin, Clinical Professor, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: S61020
Record Dates: First submitted 2020-11-24; First posted 2021-01-26 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Parkinson Disease; Essential Tremor
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Intervention Model Description: Randomized, crossover, double-blinded design
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blinded design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard clinical pulse shape (Active Comparator): Standard clinical pulse shape as used in clinical practice (cathodic stimulation).
  Interventions: Device: Boston Scientific: Study tool computer
- Complex pulse shape (Experimental): Complex pulse shape (i.e. biphasic pulse shape anode first, biphasic pulse shape cathode first, hyperpolarizing pre-pulse or depolarizing pre-pulse)
  Interventions: Device: Boston Scientific: Study tool computer

INTERVENTIONS:
Device: Boston Scientific: Study tool computer — compare clinical outcome measurements of complex pulse shapes to standard clinical pulse shape

SUMMARY:
Parkinson's disease and essential tremor are chronic movement disorders for which there is no cure. When medication is no longer effective, deep brain stimulation (DBS) is recommended. Standard DBS is a neuromodulation method that uses a simple monophasic pulse, delivered from an electrode to stimulate neurons in a target brain area. This monophasic pulse spreads out from the electrode creating a broad, electric field that stimulates a large neural population. This can often effectively reduce motor symptoms. However, many DBS patients experience side effects - caused by stimulation of non-target neurons - and suboptimal symptom control - caused by inadequate stimulation of the correct neural target. The ability to carefully manipulate the stimulating electric field to target specific neural subpopulations could solve these problems and improve patient outcomes. The use of complex pulse shapes, specifically biphasic pulses and asymmetric pre-pulses, can control the temporal properties of the stimulation field. Evidence suggests that temporal manipulations of the stimulation field can exploit biophysical differences in neurons to target specific subpopulations. Therefore, our aim is to evaluate the effectiveness of complex pulse shapes to reduce side effects and improve symptom control in DBS movement patients.

DETAILED DESCRIPTION:
The study had three stages. In the first stage, a wide range of investigatory pulse shapes in a small number of patients. The effect of the pulses on the therapeutic window will be assessed.

Stage 2 will perform a short-term chronic evaluation in a larger number of patients of the complex pulse shape selected as most interesting from stage 1.

* ET patients will first be assessed after 3 hours of the cathodic or complex pulse (double-blind design).
* PD patients will only be assessed after 1 week of each pulse.

Stage 3 will then focus on long-term evaluation (upto 2 years). Outcomes: see stage 2.

ELIGIBILITY:
Inclusion Criteria for PD:

* Diagnosis of idiopathic Parkinson's disease where the diagnosis was made by a Movement Disorder Specialist according to the MDS criteria of 2015, with a Hoehn and Yahr scale (H&Y) of at least 2 (bilateral involvement).
* Onset of the symptoms more than five years ago.
* MDS-UPDRS-III score of ≥30 without medication or DBS.
* Electrodes are implanted in target area STN.

Inclusion Criteria for ET:

* Patient is diagnosed with essential tremor by a Movement Disorder Specialist.
* Diagnosis since more than 3 years.
* Patient has a disabling medical-refractory upper extremity tremor without medication or DBS.
* Patient has a postural or kinetic tremor severity score of at least 3 out of 4 in the extremity intended for treatment on the Fahn-Tolosa-Marin Clinical Rating Scale for Tremor without medication or DBS.
* Electrodes are implanted in target area VIM.

General Inclusion Criteria:

* Post-op the implanted electrodes pass an integrity check, i.e. no open or shorted electrodes.
* Stable medications
* Lack of dementia or depression.
* Patient is willing and able to comply with all visits and study related procedures
* Patient understands the study requirements and the treatment procedures and provides written informed consent before any study-specific tests or procedures are performed.
* Patient can tolerate at least 12 hours OFF medication and per clinical judgement be able to perform all study related procedures

Exclusion Criteria:

* Any significant psychiatric problems, including unrelated clinically significant depression.
* Any current drug or alcohol abuse.
* Any history of recurrent or unprovoked seizures.
* Have any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints, including any terminal illness with survival <12 months.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Stage 1: Therapeutic window = Amplitude at which therapeutic benefit is obtained versus amplitude at which side-effects occur, both expressed in mA (milliamperes). | Immediately after testing
  Amplitude at which therapeutic benefit is obtained versus amplitude at which side-effects occur, both expressed in mA (milliamperes).
Stage 2 ET (3 hours): tremor scores | Measured after 3 hours of stimulation
  FTM (Fahn-Tolosa-Marin) total score. Max 116 (higher score for more tremor).
Stage 2 ET (3 hours): ataxia scores | Measured after 3 hours of stimulation
  ICARS (International cooperative ataxia rating scale): total score. Max 100 (higher score for more ataxia).
Stage 2 ET (1 week): number of treatment-related adverse events as assessed by CTCAE v4.0 | During 1 week of stimulation
  Follow-up of (S)AE related to the study during that week
Stage 2 PD (1 week): number of treatment-related adverse events as assessed by CTCAE v4.0 | During 1 week of stimulation
  Follow-up of (S)AE related to the study during that week
Stage 3 ET (2 years): number of treatment-related adverse events as assessed by CTCAE v4.0 | During 2 years of stimulation
  Follow-up of (S)AE related to the study during those 2 years

SECONDARY OUTCOMES:
Stage 1: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Upto one week after the study visit of stage 1
  Follow-up of (S)AE related to the study upto 1 week after the experiment
Stage 2 ET (3 hours): Therapeutic window: Amplitude to elicit tremor arrest, amplitude to elicit ataxia, amplitude to elicit stim-induced side-effects | Immediately after testing
  Amplitude to elicit tremor arrest, amplitude to elicit ataxia, amplitude to elicit stimulation-induced side-effects (all expressed in mA)
Stage 2 ET (3 hours): tremor subscores | Measured at 1 hours, 2 hours and 3 hours after start of stimulation
  FTM (Fahn-Tolosa-Marin) subscores: items 5, 6, 11, 12 and 13 (max 48, higher score for more tremor)
Stage 2 ET (3 hours): ataxia subscores | Measured at 1 hours, 2 hours and 3 hours after start of stimulation
  ICARS (international cooperative ataxia rating scale): item 10 (max 8, higher score for more ataxia)
Stage 2 ET (3 hours): speech assessment (least dysarthria) | Measured at 1 hours, 2 hours and 3 hours after start of stimulation
  Tests: sustained phonation /a/, diadochokinesis /tatata/, text reading and spontaneous speech Outcome: which of both pulses has less dysarthria per test (either cathodic pulse, either experimental pulse)
Stage 2 ET (1 week): tremor scores and subscores | Measured after 1 week of stimulation
  FTM (Fahn-Tolosa-Marin) tremor rating scale:
  * total score (max 116, higher score for more tremor)
  * subscores: items 5, 6, 11, 12 and 13 (max 48, higher score for more tremor)
Stage 2 ET (1 week): ataxia subscores and total score | Measured after 1 week of stimulation
  ICARS (international cooperative ataxia rating scale):
  * total score: max 100, higher score for more ataxia
  * subscore: item 10 (max 8, higher score for more ataxia)
Stage 2 ET (1 week): tremor measured with Kinesia One wearable | Measured after 1 week of stimulation
  Amount of postural tremor and kinetic tremor in both hands (max 4 per side, higher score for more tremor)
Stage 2 ET (1 week): tremor time measured with Kinesia 360 | Measured during 1 week of stimulation
  Amount of tremor time measured with Kinesia 360 wearable (%, higher score for more tremor time)
Stage 2 ET (1 week): speech assessment (least dysarthria) | Measured after 1 week of stimulation
  Tests: sustained phonation /a/, diadochokinesis /tatata/, text reading and spontaneous speech Outcome: which of both pulses has less dysarthria per test (either cathodic pulse, either experimental pulse)
Stage 2 ET (1 week): cognition | Measured after 1 week of stimulation
  MoCA (Montreal Cognitive Assessment). Max 30, higher score for better cognition.
Stage 2 ET (1 week): quality-of-life | Measured after 1 week of stimulation
  QUEST (Quality-of-life in essential tremor questionnaire). Max 100%, higher score for worse quality-of-life.
Stage 2 ET (1 week): quality-of-life | Measured once daily during 1 week of stimulation
  VAS (visual analogue scale) for:
  * amount of tremor
  * discomfort due to tremor Max 10, higher scores for worse outcome.
Stage 2 PD (1 week): therapeutic window (amplitude at loss of rigidity and amplitude at stim-induced side-effects) | Immediately after testing
  Amplitude at loss of rigidity and amplitude at stimulation-induced side-effects
Stage 2 PD (1 week): assessment motor symptoms in Parkinson's | Measured after 1 week of stimulation
  MDS-UPDRS-III (Movement Disorders Society Unified Parkinson's Disease Rating Scale, part III). Max 132, higher score for more parkinsonian symptoms.
Stage 2 PD (1 week): assessment non-motor symptoms in Parkinson's | Measured after 1 week of stimulation
  NMSS (non-motor symptoms scale). Max 30, higher scores for more symptoms.
Stage 2 PD (1 week): assessment of motor symptoms in Parkinson's with Kinesia One wearable | Measured after 1 week of stimulation
  Wearable scores finger tapping and hand opening. Max 4 per item, higher scores for more symptoms.
Stage 2 PD (1 week): assessment motor symptoms in Parkinson's with Kinesia 360 wearable | Measured after 1 week of stimulation
  Wearable score amount of time that patient was bradykinetic and dyskinetic. Expressed as %, higher scores for more symptoms
Stage 2 PD (1 week): assessment of speech (least dysarthria) | Measured after 1 week of stimulation
  Tests: sustained phonation /a/, diadochokinesis /tatata/, text reading and spontaneous speech Outcome: which of both pulses has less dysarthria per test (either cathodic pulse, either experimental pulse)
Stage 2 PD (1 week): cognition | Measured after 1 week of stimulation
  MoCA (Montreal Cognitive Assessment). Max 30, higher score for better cognition.
Stage 2 PD (1 week): quality-of-life | Measured after 1 week of stimulation
  PDQ-39 (Parkinson's disease Questionnaire): 39-item questionnaire on quality-of-life.
  Expressed in %, higher score for more symptoms.
Stage 2 PD (1 week): quality-of-life | Measured once daily during 1 week of stimulation
  VAS (visual analogue scale) for:
  * amount of parkinsonian symptoms
  * discomfort due to parkinsonian symptoms Max 10, higher scores for worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Myles Mc Laughlin, Prof. Dr., Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No